CLINICAL TRIAL: NCT00189163
Title: Pioglitazone in Hepatitis C: A Randomized, Double Blind, Placebo-controlled Study
Brief Title: Pioglitazone in Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hari S. Conjeevaram, Associate Professor of Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pio-hcv-108; IRB Protocol Number: 2004-0883; GCRC Protocol Number: 2085
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Genotype 1; Insulin Resistance; Pioglitazone
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Pioglitazone (Active Comparator): 30 mg, taken orally, once per day
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Sugar pill, taken orally, once a day
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pioglitazone — 30 mg, taken orally, once per day, for 48 weeks
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo Oral Tablet — Sugar Pill, taken orally, once per day, for 48 weeks
  Arms: Placebo

SUMMARY:
The presence of insulin resistance (IR) appears to be a key factor in the development of steatosis and disease progression in patience with Hepatitis C virus (HCV) genotype-1 infections similar to levels in Non-alcoholic fatty liver disease (NAFLD). The objective of this study is to determine whether Pioglatizone, when given along with Interferon and Ribavirin, reduces insulin resistance and lowers HCV viral levels and improved response in patients who have HCV genotype-1 infection when compared to a placebo.

DETAILED DESCRIPTION:
RESEARCH PLAN:

Chronic hepatitis C is a leading cause of cirrhosis and hepatocellular carcinoma in the U.S. and is the most common cause for liver transplantation. Treatment of chronic hepatitis C remains problematic and unsatisfactory. Several factors influence the response to treatment most importantly hepatitis C virus (HCV) genotype (sustained virological response/SVR seen in 40-45% vs. 75-80% using pegylated IFN + ribavirin combination therapy genotype 1 vs. 2/3). Recently, the presence of hepatic steatosis has been shown to be an important predictor of disease progression and also response to antiviral therapy especially in patients with genotype 1 infection. The mechanisms of hepatic steatosis in HCV are multi-factorial; the presence of insulin resistance (IR) appears to be a key factor especially in genotype 1 (metabolic steatosis) similar to that seen in patients with non-alcoholic fatty liver disease (NAFLD). Whereas metabolic steatosis appears to be a factor in resistance to antiviral therapy, viral steatosis (direct viral induced as in genotype 3) is reduced in those who achieve an SVR. We recently also observed that IR is common in type 1 HCV infection even at low BMIs and is present even in the non-steatotic hepatitis C patients, suggesting a direct effect of viral infection on insulin sensitivity and that IR may precede hepatic steatosis. We hypothesize that in patients with HCV genotype 1 infection, therapy aimed at improving insulin sensitivity in conjunction with standard antiviral therapy may not only reduce the insulin resistance in hepatitis C but also improve hepatic steatosis, decrease expression of pro-inflammatory cytokines and reduce oxidative stress thereby preventing disease progression. In addition, we also hypothesize that improvement in IR and hepatic steatosis may also result in improved virological response to antiviral therapy.

This study introduces a novel concept of using the insulin sensitizing thiazolidinedione agent pioglitazone to improve insulin sensitivity, improve hepatic steatosis and possibly result in a higher rate of virological response when given in conjunction with standard antiviral therapy in treatment naïve patients with genotype 1 infection. Our main goals are to study the effect of pioglitazone on insulin sensitivity and hepatic steatosis in addition to its effect on SVR along with confirming the safety of pioglitazone in patients with hepatitis C. To our knowledge, this is the first randomized, placebo-controlled study of an insulin sensitizing agent in the treatment of patients with chronic hepatitis C. We hope that the findings in this study will shed new light into the mechanisms associated with the pathogenesis of hepatitis C and lead to new and effective treatments in the management of this very important disease.

Insulin resistance (IR), a key factor in the development of steatosis, is a common finding in patients with hepatitis C virus (HCV) infection. In patients with genotype 1 infection, IR has been noted in up to 80% of patients in some studies. In patients with non-alcoholic fatty liver disease (NAFLD) who have evidence of nonalcoholic steatohepatitis (NASH), the role of IR leading to decreased fatty acid oxidation, increased production of pro-inflammatory cytokines and increased oxidative stress had been proposed as an important mechanism leading to steatosis and subsequent liver cell injury. Recently, an association between steatosis and hepatic fibrosis has been emphasized in HCV infection, similar to that described in patients with NAFLD. While IR and hepatic steatosis are common findings in patients with HCV infection, the latter with prevalence rates of 40% to 70%, and different HCV genotypes confers distinct risks for steatosis; a greater degree of steatosis is seen in patients with genotype 3 infection compared to others. Similar to that seen in patients with NAFLD, patients infected with genotype 1 HCV show a relationship between body mass index (BMI) and risk for steatosis. However, in up to 30% of patients with HCV infection and hepatic steatosis, no other risk factors for steatosis can be identified. The investigators' preliminary data will show that even in HCV infected individuals with low BMI and no steatosis, there is IR and the risk for steatosis is increased when directly compared to NAFLD patients. Recent data also suggest that the presence of hepatic steatosis is an independent predictor of decreased response to antiviral therapy even when controlling for genotype. This is especially important in patients with type 1 infection.

The investigators hypothesize that in patients with HCV genotype 1 infection, treatment with antiviral therapy will have a partial effect on reducing insulin resistance (IR) and steatosis and this is augmented by the addition of an insulin sensitizing thiazolidinedione (TZD) agent such as pioglitazone to the treatment regimen. The investigators also hypothesize that the rate of sustained virological response (SVR) will be higher in the antiviral regimen + pioglitazone treated group compared to patients receiving antiviral therapy alone.

The investigators' specific aims are the following:

1. To assess the improvement in insulin sensitivity in patients with treatment naïve genotype 1 chronic hepatitis C treated with standard antiviral therapy + pioglitazone or placebo
2. To assess the improvement in hepatic steatosis in patients with treatment naïve genotype 1 chronic hepatitis C after treatment with standard antiviral therapy + pioglitazone or placebo
3. To assess the rates of sustained virological response (SVR) among patients with treatment naïve genotype 1 chronic hepatitis C treated with standard antiviral therapy + pioglitazone compared to standard antiviral therapy + placebo

CLINICAL STUDY DESIGN AND METHODS

Overview:

This is a randomized, double-blind, placebo-controlled study of pioglitazone given in combination with standard antiviral therapy for the treatment of genotype 1 infected hepatitis C patients who are treatment naïve. We will determine the rates of improvement in homeostasis model assessment of insulin resistance (HOMA-IR) and hepatic steatosis after 48 weeks of therapy compared to baseline along with determining the rate of SVR in the two treatment groups. In addition, we will also assess the safety of pioglitazone in patients with chronic hepatitis C infection.

All eligible patients will have undergone a percutaneous liver biopsy within 6 months of enrollment to assess the severity of hepatitis C, steatosis and features of steatohepatitis by the study pathologist. A period of 6 months prior to enrollment was selected in order to have a more recent representation of the degree of steatosis and histologic severity of hepatitis C as the effect of therapy on these histologic features is one of the important aims in this study. A HOMA index value of > 2.0 was selected to define IR in this study (see below: Inclusion criteria) as this value is considered abnormal and indicative of decreased insulin sensitivity. Histological severity of chronic hepatitis C will be done using the modified histological activity index (HAI) scoring system by Ishak for grading and staging chronic viral hepatitis and that for steatosis and steatohepatitis will be done using the scoring system that is currently being used in the NIH-funded Virahep-C study, which the PI is currently a member.

We currently have an IRB approved protocol at the University of Michigan to collect a sample of liver tissue at the time of liver biopsy in all patients with hepatitis C and NAFLD to study fat gene expression. We will collect samples on patients being considered for this study who are undergoing a liver biopsy at initial evaluation. We will also collect similar samples at the time of repeat liver biopsies in this study. This will give us a unique opportunity to study the effect of pioglitazone on fat-related gene expression and its relationship to responses being studied in this study (changes in IR and steatosis and virological response to therapy).

Given that this is a pilot study of pioglitazone in patients with hepatitis C and the potential hepatotoxicity of this drug in hepatitis C is not well known due to limited available data, we plan to enroll treatment-naïve patients with evidence of at least some fibrosis on liver biopsy (a minimum Ishak fibrosis score of 1) although we do not have any reason to expect any significant drug induced liver injury with this drug. Patients with evidence of cirrhosis on liver biopsy (Ishak fibrosis score 5 and 6) will be excluded since cirrhosis itself can be associated with IR and thereby bias the findings. Although we do not expect to see any increased hepatotoxicity due to pioglitazone in patients with hepatitis C in general, whether cirrhosis increases potential risk is unknown at this time.

Similarly, we also plan to exclude patients with known diabetes mellitus (DM) to minimize any bias especially since interferon therapy itself can affect glucose tolerance and may lead to difficult control in patients with pre-existing diabetes. In our hepatitis C patient population, although prevalence of DM is less than 15%, the addition of diabetic patients may also confound the analysis unless we stratify randomization based on presence or absence of DM and since this is a pilot study with a limited sample size, we decided to exclude diabetics. Another factor would be correcting the influence of glucose controlling agents on insulin sensitivity during the study.

All eligible patients who are interested in the study will be invited to come to the GCRC at regular intervals for study assessment. During these visits, a brief physical examination will be performed and blood will be collected and stored for future research purposes. The current standard treatment for chronic hepatitis C patients with genotype 1 infection is a combination of pegylated interferon and ribavirin for 48 weeks. Treatment response is defined as follows:

* Sustained Virological Responder (SVR) - undetectable HCV RNA in serum during therapy and at 24 weeks follow-up;
* Relapser - undetectable HCV RNA in serum during and end of treatment and reappearance of RNA once therapy is stopped; we expect less than 15% of initial responders to relapse after stopping treatment;
* Non-Responder - presence of HCV RNA in serum at the end of therapy and during follow-up.

Although patients with genotype 1 who have detectable HCV RNA at 24 weeks of therapy are usually labeled as non-responders and treatment is stopped in clinical practice, all patients in this study will complete 48 weeks of treatment unless the regimen has to be stopped due to side effects or patient preference. This is because of potential beneficial effects of therapy (addition of pioglitazone to antiviral therapy) on IR and hepatic steatosis and possibly even fibrosis even among viral non-responders when treated for 48 weeks.

Once treatment is completed, all patients will be invited to come to GCRC 12 weeks following the end of treatment to undergo a repeat liver biopsy. Total follow-up once treatment is stopped will be 24 weeks in all patients.

Patient Population:

All eligible adult patients with compensated liver disease due to chronic infection with HCV and genotype 1 infection who are treatment naïve will be enrolled into the study. All racial and ethnic groups will be recruited into this study. Patients with cirrhosis and decompensated liver disease and any patient, in whom a liver biopsy is contraindicated, will be excluded. Race (African American/Black or non-Hispanic white or other) will be assigned based on the information given by the patient. It reflects the individual's recognition in the community. This assignment of race/ethnicity will be similar to that practiced by governmental agencies including the U.S. Census Bureau and the Center for Disease Control. All patients will sign an IRB approved HIPAA compliant consent form before enrolling into the study.

ELIGIBILITY:
Inclusion Criteria:

* All eligible adult patients with compensated liver disease due to chronic infection with HCV and genotype 1 infection who are treatment naïve will be enrolled into the study.
* All racial and ethnic groups will be recruited into this study.
* Males and females: age > 18 years
* Chronic hepatitis C: history of serum positive for HCV antibody (anti-HCV) and HCV RNA. Patients should have evidence of chronic hepatitis with a minimum fibrosis score of 1 on liver biopsy done within 6 months of enrollment.
* Insulin resistance based on HOMA index value (HOMA-IR) of > 2.0 during screening. HOMA-IR is a well recognized and validated index of insulin resistance in both non-diabetic and diabetic populations and has been shown to have a good correlation with 'clamp' techniques that are intensive. HOMA is also used routinely to assess longitudinal changes including assessment of the effects of treatment. In general, a HOMA-IR value of > 1.5 is considered abnormal based on repeat testing measurements performed by both HOMA assessment and by euglycemic clamp technique and is considered representative of decreased insulin sensitivity. Although insulin secretion is pulsatile, the correlation between HOMA computed from repeat sampling (using a mean of three samples taken at 5-minute intervals to compute HOMA) and the value obtained from a single basal sample to determine insulin sensitivity has been shown to be near perfect even in patients with type 2 diabetes (r = 0.99, p < 0.0001). The investigators will use a HOMA-IR value of > 2.0 as part of the inclusion criteria in this study.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Hepatitis C patients who underwent previous therapy for their liver disease
* Genotype other than type 1
* Histological evidence of cirrhosis or confirmed hepatocellular carcinoma (HCC)
* Patients with cirrhosis and decompensated liver disease and any patient, in whom a liver biopsy is contraindicated, will be excluded.
* Evidence of other causes of chronic liver disease
* Diabetes mellitus
* New York Heart Association (NYHA) functional classification for cardiac disease: class III and IV patients
* Human immunodeficiency virus (HIV) antibody positive
* Patients with solid organ transplants
* Pregnancy or breast feeding
* Participation in any other clinical trial within 90 days of entry into this trial.
* Unwilling to consent to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Virologic Response | 72 weeks
  Measuring HCV RNA in serum (detectable or undetectable)

SECONDARY OUTCOMES:
Change from Baseline in Insulin Sensitivity | 72 weeks
  HOMA Index
Change from Baseline in Histology | 60 weeks
  ISHAK Score

CONTACTS AND LOCATIONS:
Overall Officials: Hari S Conjeevaram, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States